

### Study consent form

Official study title: The effect of consuming grass finished lamb meat on omega-3 blood response among healthy consumers

NCT number: 19.08v2

Date: 22/03/2019



### **Consent Form**

# Project title: The effect of consuming grass finished lamb meat on omega-3 blood response among healthy consumers

#### Please initial box

| 1. | I confirm that I have been given and have read and understand the Information Leaflet for the above study. I have had the opportunity to ask, and receive answers to any questions I may have had. | | | [ | ] |
|---|---|---|---|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason. | | | [ | ] |
| 3. | I agree to take part in the above study, inclusive of the procedures mentioned in the Information Leaflet (completion of questionnaire, blood sampling, blood pressure and body mass index measures) | | | [ | ] |
| 4. | I understand that my participation or non-participation will not affect my career progression, my medical care or my legal rights being affected in anyway. | | | | ] |
| 5. | I understand all data will be treated securely as described by the new EU General Data Protection Regulation and stored appropriately as required by the University. | | | [ | ] |
| 6. | I understand that I will not be identifiable in any data published in relation to this project. | | | [ | ] |
| l agre | e to take part in this project | | | | |
| Name of Participant | | Date | Signature | | |
| | of Person taking consent<br>erent from Researcher) | Date | Signature | | |
| Name | of Researcher | Date | Signature | | |

## Consent form version 19.08v2 22/03/2019

Name of Researcher: Lynda Perkins (PhD student) Email: I.perkins@qub.ac.uk/lambstudy@qub.ac.uk

Phone number: 07980946197

Name of supervisor: Professor Nigel Scollan

Email: Nigel.Scollan@qub.ac.uk Phone number: +44 (0)28 9097 6549

Name of supervisor: Dr. Anne Nugent

Email: A.Nugent@qub.ac.uk

Phone number: +44 (0)28 9097 4167

Name of supervisor: Professor Jayne Woodside

Email: j.woodside@qub.ac.uk

Phone number: +44 (0)28 9097 8942